CLINICAL TRIAL: NCT05697302
Title: The Effect of Training and Follow-up Given to Mothers with 15 Day-4 Month-old Babies According to the Health Promotion Model on Relactation Success: a Randomized Controlled Study
Brief Title: The Effect of Training and Follow-up Given According to the Health Promotion Model on Relactation Success
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Ayşe Daştan Yılmaz, Principal Investigator, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TDK-2023-10842
Record Dates: First submitted 2023-01-02; First posted 2023-01-25 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Breastfeeding
Keywords: Health Promotion Model; Relactation; Lactation
MeSH Terms: conditions — Breast Feeding | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Relactation (Experimental)
  Interventions: Behavioral: Education; Behavioral: Follow-up
- Control (Active Comparator)
  Interventions: Behavioral: Follow-up; Behavioral: Referral to Lactation and Relactation Polyclinic

INTERVENTIONS:
Behavioral: Education — Interviews will be held twice a week in the first two weeks of the first month, once a week in the following weeks, and once every two weeks in the second month, 8 times in a total of 2 months. The number of 8 interviews planned in the research may increase specifically for the situation of the mother and the baby. Interviews will be held at the mothers' homes or at the Family Health Center. An individualized message will be sent to mothers, two days a week, in accordance with their mobile communication tool, relactation needs. In addition, if the mothers request, they can call the researcher via mobile communication via video or voice and receive live support regarding their questions and questions.
  Arms: Relactation
Behavioral: Follow-up — Among the data collection forms, LATCH-Breastfeeding Diagnostic Scale and IMDAT-The Baby's Breastmilk Scoring System will be applied at each interview, and the Breastfeeding Self-Efficacy Scale and Breastfeeding Motivation Scale will be applied at the first interview, at the end of the 1st month and at the end of the 2nd month. Mother interviews will be held in their homes or at the Family Health Center (whichever they prefer). At each meeting, an appointment schedule will be made for the next meeting and this information will be shared with the mothers in writing.
Behavioral: Referral to Lactation and Relactation Polyclinic — Due to the nature of the research, mothers in the control group will not be given any training, and they will be referred to the Lactation and Relaxation Polyclinic in Erzincan Mengücek Gazi Training and Research Hospital.
  Arms: Control

SUMMARY:
The process of restarting or increasing lactation in a mother who wants to breastfeed her baby again after the termination of breastfeeding or decrease in lactation is called relactation. The research type was planned as a pretest-posttest randomized controlled experimental study. The research will be carried out between January 2023 and December 2023, with mothers in need of relactation identified in Erzincan Binali Yıldırım University Mengücek Gazi Training and Research Hospital and 7 Family Health Centers in Erzincan city center. The study will be face-to-face, twice a week in the first two weeks of the 1st month, once a week in the other weeks, and once every two weeks in the 2nd month, in a total of 2 months, and will consist of 8 interviews. The number of these meetings may increase depending on the situation of the mother and the baby. Interviews will be held at mothers' homes or at FHCs (whichever they prefer). During the research, based on the SGM, training on the importance of breast milk and breastfeeding, its benefits and relactation techniques, written and visual training materials containing these topics, online messages and online live support by calling the researcher by video or audio when requested, and the breastfeeding process will be supported. The sample will consist of 70 mothers, 35 of whom are in the intervention group and 35 of them are in the control group, who meet the research criteria. In data collection, the World Health Organization (WHO) Simple Routine Evaluation and Breastfeeding Assistance form, Personal Information Form, Breastfeeding Self-Efficacy Scale (EÖYÖ), Breastfeeding Diagnostic Measurement Tool (LATCH) and IMDAT- Scoring System for the Amount of Breastmilk Ingested by the Baby, Breastfeeding Motivation Scale (EMO) and VAS satisfaction scale will be used. Study; The aim of this study was to determine the effect of the education and follow-up given to mothers who need help with relactation on the success of relaxation. The data will be evaluated with the IBM SPSS (Statistical Package for Social Sciences) 22.0 package program. Frequency and percentage will be used in the analysis of the data. In addition, necessary analyzes will be made after testing whether the data obtained comply with the normal distribution. P<0.05 will be used as the 95% confidence interval and significance level in the results.

ELIGIBILITY:
Inclusion Criteria:

* Can read and write Turkish and has no speech impediment,
* Being between the ages of 18-45 and having given birth for the first time,
* Mother and baby not having any health problems that would prevent breastfeeding (medications used in cancer treatment in the mother, some epilepsy medications, psychotherapy medications, migraine medications, Parkinson's medications, some painkillers, radioactive iodine use, active tuberculosis, HIV infection; congenital anomaly, galactosemia disease, phenylketonuria disease, congenital metabolic disease such as urea cycle enzyme defect),
* Not breastfeeding for at least 2 weeks and at most 8 weeks (for mothers who have never breastfed)
* Decreased milk supply that causes babies to be fed with formula for more than 2 weeks (for mothers with low milk supply),
* Having breastfeeding problems that cause decreased milk supply (breast refusal, incorrect breastfeeding techniques, breast abscess… starting work early…). •Separation of the baby or mother due to hospitalization, A mother who is formula feeding her baby changes her mind,
* No use of drugs that will affect the amount of milk (galactagogues such as metoclopramide, domperidone),
* The mother can be reached by phone,
* The baby is at least 15 days old and at most 4 months old.

Exclusion Criteria:

* Adopted/non-biological babies,
* Any health condition that would prevent breastfeeding or breastfeeding in the mother or baby (medications used in cancer treatment, some epilepsy medications, psychotherapeutic medications, migraine medications, Parkinson's medications, some painkillers, radioactive iodine use, active tuberculosis, HIV infection in the mother; congenital anomaly in the baby, galactosemia disease, phenylketonuria disease, congenital metabolic disease such as urea cycle enzyme defect), Use of medication that would affect milk quantity (galactagogues such as metoclopramide, domperidone)
* Women participating in another study on breastfeeding during the study period will not be included in the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2025-01-04 (Actual)

PRIMARY OUTCOMES:
Determination of mothers' breastfeeding self-efficacy level | 4 months
  The personal information of the mothers who agreed to participate in the study will be recorded, and the breastfeeding self-efficacy level of the mothers will be determined. For this purpose, the Breastfeeding Self-Efficacy Scale will be used. The scale consists of 14 items assessing breastfeeding self-efficacy. The scale is in a 5-point Likert type and the items of the scale are evaluated by grading from 1 = 'I am not sure at all' to 5 = 'I am always sure'. The lowest score that can be obtained from the scale is 14, and the highest score is 70; A higher score means higher breastfeeding self-efficacy.
Relactation success | 4 months
  As a criterion to show that relactation is provided, the daily amount of fluid that the baby should take in the form of 150 ml / kg / day.
  The amount of liquid in one meal obtained by dividing the number of feedings will be based on. According to the realization of the relactation,, it will be evaluated as partial (relactation occurs but the continuation of formula feeding with breastfeeding), complete (relactation occurs and the baby is fed only through breastfeeding) or unsuccessful (inability to provide relactation despite all the applications), and the relactation response is considered positive in the following cases. will be: tingling sensation in the breast during breastfeeding; appearance of milk in manual milking; reduction in the daily amount of supplemental milk given to the baby; and infant weight gain. Once a positive response is observed, additional milk supplements will be gradually reduced as breast milk secretion increases.
Determination of mothers' breastfeeding motivation | 4 months
  The personal information of the mothers who accepted to participate in the study will be recorded and the breastfeeding motivation levels of the mothers will be determined. For this purpose, the Breastfeeding Motivation Scale will be used. The scale is in 4-point Likert type and is scored between 1=Strongly Disagree and 4=Strongly Agree for each item. Each item is scored between 1-4. Accordingly, the lowest score that can be obtained from the scale is 23 in primiparous mothers, 24 in multiparous mothers, the highest score is 92 in primiparous mothers and 96 in multiparous mothers. The fact that the values obtained as a result of the study are close to the highest scores indicates that the motivation for breastfeeding is high.
Determination of amount of breast milk the baby receives. | 4 months
  The personal information of the mothers who agreed to participate in the study will be recorded, and the amount of breast milk the baby receives will be determined. For this purpose, the Scoring System for the Amount of Breastmilk Taken by the Baby will be used. The form consists of 5 sections: the weight of the babies, their satisfaction, the frequency and characteristics of urinating and defecation, and the condition of the mother's breasts. With the form, the features of each situation are evaluated as 0, 1, 2 points, and the maximum total score that can be obtained is 10. A score of 8-10 is considered the best breast milk intake, and a score of 0-7 is considered insufficient. This scoring system will be applied in every follow-up, and additional food/food intake management of the baby will be done in line with the information in possible relactation success.
Breastfeeding diagnosis of mothers | 4 months
  The personal information of the mothers who agreed to participate in the study will be recorded, and breastfeeding diagnosis of mothers will be made. For this purpose, the Breastfeeding Diagnostic Scale will be used. This measurement tool consists of five evaluation criteria, which is a combination of the first letters of the English equivalent of these criteria. LATCH's evaluation criteria; L-Latch on breast, A-Audible swallowing, T-Type of nipple, C-Comfort nipple, H-Hold. Each item is evaluated between 0-2 points. The total score that can be taken from the scale is 10.

SECONDARY OUTCOMES:
Levels of satisfaction with the education and follow-up of mothers | 4 months
  "Vissuel Analog Scale (VAS)" will be used to determine the satisfaction of mothers in the intervention group with the nursing care provided to them such as SGM-based education, monitoring, relaxation practices, telephone support, education and monitoring at home, and education and monitoring in FHC. In the scale, mothers will be asked to express their satisfaction level with numbers as "0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10".

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe DAŞTAN YILMAZ, Principal Investigator — Erzincan Binali Yildirim Universitesi; Kıymet YEŞİLÇİÇEK ÇALIK, Principal Investigator — Karadeniz Teknik University
Locations (1):
- Karadeniz Teknik Üniversitesi, Trabzon, Turkey (Türkiye)